CLINICAL TRIAL: NCT04846491
Title: A Multi-center, Randomized, Blinded Study to Evaluate the Efficacy and Safety of Peginterferon Alfa-2b Injection Combined With Tenofovir Disoproxil Fumarate Tablets in Patients With Chronic Hepatitis B
Brief Title: A Study of Peginterferon Alfa-2b Combined With TDF in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TB1901IFN
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-08

CONDITIONS: Chronic Hepatitis B
Keywords: peginterferon alfa-2b injection; interferon alfa; nucleos(t)ide; NUCs; NAs; chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nucleot(s)ide-treated patients-Experimental Group 1 (Experimental)
  Interventions: Drug: Peginterferon alfa-2b injection
- Nucleot(s)ide-treated patients-Experimental Group 2 (Experimental)
  Interventions: Drug: Peginterferon alfa-2b injection
- Nucleot(s)ide-treated patients-Control Group (Active Comparator)
  Interventions: Drug: TDF
- Treatment Naive Group (Other)
  Interventions: Drug: Peginterferon alfa-2b injection

INTERVENTIONS:
Drug: Peginterferon alfa-2b injection — Peginterferon alfa-2b injection (high dose) will be weekly subcutaneous injected for 8 weeks and then stop for 4 weeks, 12 week a cycle, up to 12 cycles (144 weeks) at most. TDF will be taken orally during the whole treatment period. And then followed for 24 weeks after treatment.
  Arms: Nucleot(s)ide-treated patients-Experimental Group 1
Drug: Peginterferon alfa-2b injection — Peginterferon alfa-2b injection (low dose) will be weekly subcutaneous injected for 8 weeks and then stop for 4 weeks, 12 week a cycle, up to 12 cycles (144 weeks) at most. TDF will be taken orally during the whole treatment period. And then followed for 24 weeks after treatment.
  Arms: Nucleot(s)ide-treated patients-Experimental Group 2
Drug: TDF — Patients will take TDF orally for the first 48 weeks, and then one can choose to continue the single-TDF treatment up to 144 weeks, or may choose to change to receive peginterferon alfa-2b combined TDF therapy for the later 96 weeks, peginterferon alfa-2b will be weekly subcutaneous injected for 8 weeks and then stop for 4 weeks, 12 weeks a cycle. And then followed for 24 weeks after treatment.
  Arms: Nucleot(s)ide-treated patients-Control Group
Drug: Peginterferon alfa-2b injection — Peginterferon alfa-2b injection will be weekly subcutaneous injected for 8 weeks and then stop for 4 weeks, 12 week a cycle, up to 12 cycles (144 weeks) at most. TDF will be taken orally during the whole treatment period. And then followed for 24 weeks after treatment.
  Arms: Treatment Naive Group

SUMMARY:
Current clinical practices has shown promising prospects of the therapy strategy of interferon combined with nucleos(t)ides in patients with chronic hepatitis B, but the safety and efficacy has not been fully studied. This study is aimed to exploit the safety and efficacy of the study drug, Peginterferon alfa-2b injection, with nucleos(t)ide (NAs), tenofovir disoproxil fumarate tablets (TDF), in the patients with hepatitis B, who has previously treated with nucleos(t)ides and who are treatment naïve.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign the informed consent form voluntarily.
* Age between 18 and 65 years (including 18 and 65), no gender limit.
* HBsAg-positive for at least 6 months or other evidence supporting chronic infection with hepatitis B virus.
* HBsAg positive at screening.
* For NAs treated patients: Who should have continuously taken NAs for at least 9 months prior to screening, and are currently receiving the NAs. Simultaneously, the patients should have achieved the following criteria: HBsAg<1500IU/mL, HBV DNA<100IU/ml, HBeAg<10s/co at screening.
* For treatment naive patients: HBV DNA≥1×10^4IU/ml, and 2×ULN (upper limit of normal) ≤ALT≤10×ULN at screening.
* Pregnancy test of female of childbearing must be negative within 24 hours before the first medication, and the subjects (male and female) should take effective contraceptive measures during the whole study period.

Exclusion Criteria:

* Women who are pregnant, breastfeeding or planning to pregnant during the study period.
* Subjects with neuropsychiatric diseases and/or neuropsychiatric family history, especially depression, anxiety, or mania schizophrenia.
* Co-infected with Hepatitis A, Hepatitis C, Hepatitis D, Hepatitis E, or HIV.
* Chronic hepatitis other than hepatitis B, e.g. alcoholic hepatitis, drugs-induced hepatitis, or autoimmune hepatitis, etc.
* Moderate to severe steatohepatitis.
* Evidence of acute severe hepatitis, e.g. ALT>10×ULN, significantly increasing in ALT accompanied by elevated bilirubin, etc.
* Evidence of liver decompensation, e.g. total bilirubin higher than 2×ULN, albumin lower than 35g/L, prothrombin time is 3 seconds longer than the upper limit of normal, prothrombin activity lower than 60%, or history of decompensated liver cirrhosis, etc.
* Evidence of hepatocellular carcinoma, or AFP>1×ULN.
* Significant kidney diseases, including acute nephritis, chronic nephritis, renal insufficiency, nephrotic syndrome, etc. or serum creatinine higher than upper limit of normal.
* Neutrophil count less than 1.5×10^9/L, or platelet count less than 90×10^9/L at screening.
* Serum phosphorus lower than 0.8mmol/L.
* Antinuclear antibody (ANA) exceeds 1:100.
* Autoimmune disease, including psoriasis, systemic lupus erythematosus, etc.
* Subjects with endocrine system disease, including thyroid, Diabetes mellitus, etc.
* Poorly controlled hypertension (blood pressure ≥140/90 mmHg).
* Subjects with severe heart disease, especially those with unstable angina or poorly controlled heart disease within 6 months prior to screening.
* Severe retinopathy or any other severe diseases in the eyes.
* Subject who had ever received organ transplants or are planning to receive organ transplant.
* For NAs-treated patients: who have received standard treatment of interferon products within 6 months prior to screening .
* For treatment naive patients: who have ever received standard treatment of interferon products, or who have ever received NAs within 6 months prior to screening.
* Subject who are allergic to interferon, tenofovir, or any excipients, or meet any of the contraindications described in the drug instructions.
* Subjects who participated in any other interventional trials within 3 months prior to screening, or with any other conditions which in the opinion of the investigator precluding enrollment from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBsAg negative. | 24 weeks post treatment.

SECONDARY OUTCOMES:
Changes of HBsAg level from baseline. | up to 168 weeks.
Proportion of patients with HBsAg seroconversion. | up to 168 weeks.
Proportion of patients with HBeAg negative. | up to 168 weeks
Proportion of patients with HBeAg seroconversion. | up to 168 weeks.
Changes of HBeAg level from baseline. | up to 168 weeks.
Proportion of patients with HBV DNA undetectable. | up to 168 weeks.
Changes of HBV DNA level from baseline. | up to 168 weeks.
Proportion of patients with ALT normalization. | up to 168 weeks.
Proportion of patients with liver fibrosis. | up to 168 weeks.
Proportion of patients with liver cirrhosis. | up to 168 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Ph.D, Principal Investigator — Peking University First Hospital
Locations (33):
- China (33):
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - The fifth medical center of PLA General Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Public Health Clinical Center of Chengdu, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Mengchao Hepatobiliary Hosipital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The Ninth Hospital of the Joint Logistic Support Force of the Chinese People's Liberation Army, Fuzhou
  - Guangzhou Eighth People's Hospital, Guangzhou
  - The Third Affiliated Hospital,SUN YAT-SEN University, Guangzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Nanjing Drum Tower Hospital/The First Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Huashan Hospital affiliated to Fudan University, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The Sixth People's Hospital of Shenyang, Shenyang
  - Peiking University Shenzhen Hospital, Shenzhen
  - The Third People's Hospital of shenzhen, Shenzhen
  - The First Hospital of Shanxi Medical University, Taiyuan
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin
  - Tianjin Third Central Hospital, Tianjin
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Traditional Chinese Medicine hospital of Xinjiang Uygur Autonomous Region, Ürümqi
  - Tongji Hospital/Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - Tangdu Hospital, Xi'an
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen
  - Yanbian University Hospital/Yanbian Hospital, Yanbian
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No